CLINICAL TRIAL: NCT03833245
Title: Optimizing Pregnancy and Treatment Interventions for Moms 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jerry Cochran, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 116398
Record Dates: First submitted 2019-01-28; First posted 2019-02-06 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy, High Risk; Opioid-Related Disorders; Pregnancy Related
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The standard care condition includes brief case management and referral. The brief case management involves the participant speaking to a hospital social worker who conducts a patient needs assessment in the areas of behavioral health and social services. All patients will be referred to MAT and any identified behavioral health or social service needs.
- Patient Navigation (Experimental): The prenatal portion of the intervention includes 10 sessions delivered within approximately 14 weeks. The postnatal portion of the intervention will be delivered as 4 sessions over 8 weeks. Women who complete the intervention before delivery will receive regular calls/texts until delivery wherein the navigator will encourage and reinforce abstinence and treatment retention.
  Interventions: Behavioral: Patient Navigation

INTERVENTIONS:
Behavioral: Patient Navigation — The patient navigation (PN) intervention will initiate following participant recruitment. It is important to note that PN sessions do not strictly coincide with specific weeks of pregnancy since the women can be recruited up to ≤25 weeks of gestation. The prenatal portion of the intervention includes 10 sessions delivered within approximately 14 weeks. The postnatal portion of the intervention will be delivered as 4 sessions over 8 weeks. Women who complete the intervention before delivery will receive regular calls/texts until delivery wherein the navigator will encourage and reinforce abstinence and treatment retention. All contact will be reported by staff in a patient contact log developed for the study that will be used to quantify level of patient contact.
  Arms: Patient Navigation

SUMMARY:
The US opioid epidemic continues to result in serious health consequences for pregnant and postpartum women. In the US from 2007 to 2012, an average of 21,000 pregnant women each year reported past month opioid misuse. This study aims to provide rapid and targeted primary prevention activities aimed at assisting pregnant women with opioid use disorder (OUD) to become linked to and retained in treatment in order to reduce harms to them (including overdose) and their offspring.

DETAILED DESCRIPTION:
Age adjusted rates for overdose among women in the US increased more than six-fold from 1.4 in 1999 to 8.5 in 2016. Examining Pennsylvania (PA) and Utah (UT; the states where recruitment will happen in this study), these states have some of the highest rates of overdose among women compared to other US states. Specifically, PA's overdose rate among women surpassed the national average in 2016, and rates of overdose death in UT among women have ranged 2-9 times higher than the national rate between 2009 to 2016. Both PA and Utah are among the states with the highest opioid prescribing to pregnant women, with Utah being the highest in the nation (41.6%). Prenatal opioid use disorder (OUD) in the US has brought serious health consequences for mother and infant-including preterm delivery, low birth weight, NAS, and poor breastfeeding, and includes substantial expenditures of health care resources. Chances for HIV (OR=20.3, 95% CI = 13.8-29.7) and hepatitis C virus (OR=150.2. 95% CI = 120.9-186.6) infection among women with OUD are markedly higher than for those without OUD. Pregnant women with OUD have high rates of psychiatric illnesses, such as depression and anxiety, and other substance use disorders (SUDs), with particularly high rates of smoking (>80%). Neonatal abstinence syndrome (NAS), an opioid withdrawal syndrome among neonates, has also increased substantially from 3.4/1000 births in 2009 to 5.8/1000 births in 2012. Poly-substance use among pregnant women with OUD has also been associated with higher levels of needed medications to treat NAS and longer duration of NAS treatment. Smoking combined with opioid use during pregnancy has likewise been related to longer duration of NAS treatment, greater NAS severity, and higher levels of medication needed to treat NAS symptomology. Any prenatal opioid use also has been associated with birth defects, including neural tube defects, conoventricular septal defects, atrioventricular septal defects, hypoplastic left heart syndrome, and gastroschisis. Compared with women without any SUDs, children born to mothers with OUD or OUD plus other SUDs also have been documented to have lower cognitive functioning as they mature. Problems resulting from illicit and prescription OUD also result in significant social issues. Pregnant women with OUD have been observed to have financial and housing instability, challenges related to employment, and involvement with the legal system.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* English speaking
* Pregnant women (pregnancy status verified by gestational age >6 weeks from last menstrual period confirmed by ultrasound)
* OUD verified by examination of medical records for an OUD diagnosis, urine toxicology, and the Diagnostic and Statistical Manual of Mental Disorders (DSM) Checklist (modified from the DSM-IV to confirm current diagnosis for substance use disorders)
* Plan to carry their babies to delivery verified by patient self report

Participant Exclusion Criteria

* Experienced a psychotic or a manic episode in the last 30 days documented in their medical record
* Beyond the 25th week of gestation
* Cannot provide collateral contact information of 2 persons,
* Cannot provide a reliable phone number,
* Plan to move from the area within 2 months of their delivery will or 6 months after not be included in the study
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.
* Other factors that would cause harm or increased risk to the participant or close contacts, or preclude the participant's full adherence with or completion of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Cochran, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cochran G, Smid MC, Krans EE, Yu Z, Carlston K, White A, Abdulla W, Baylis J, Charron E, Okifugi A, Gordon AJ, Lundahl B, Silipigni J, Seliski N, Haaland B, Tarter R. Patient navigation for pregnant individuals with opioid use disorder: Results of a randomized multi-site pilot trial. Addiction. 2024 Mar;119(3):544-556. doi: 10.1111/add.16364. Epub 2023 Oct 20. PMID 37859587
- [Derived] Charles JE, Baylis J, Smid MC, Cochran G. Nonfatal Overdoses Among Pregnant Individuals With Opioid Use Disorder. Obstet Gynecol. 2023 May 1;141(5):961-963. doi: 10.1097/AOG.0000000000005129. Epub 2023 Apr 5. PMID 37103536
- [Derived] Bryan MA, Mallik D, Cochran G, Lundahl B. Mindfulness and Savoring: A Commentary on Savoring Strategies and Their Implications for Addiction Treatment. Subst Use Misuse. 2022;57(5):822-826. doi: 10.1080/10826084.2022.2046090. Epub 2022 Mar 10. PMID 35349380
- [Derived] Cochran G, Smid MC, Krans EE, Bryan MA, Gordon AJ, Lundahl B, Silipigni J, Haaland B, Tarter R. A pilot multisite study of patient navigation for pregnant women with opioid use disorder. Contemp Clin Trials. 2019 Dec;87:105888. doi: 10.1016/j.cct.2019.105888. Epub 2019 Nov 12. PMID 31731006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Patient Navigation
Started | 49 | 53
Completed | 49 | 52
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: The standard care condition includes brief case management and referral. The brief case management involves the participant speaking to a hospital social worker who conducts a patient needs assessment in the areas of behavioral health and social services. All patients will be referred to MAT and any identified behavioral health or social service needs.
- Total: Total of all reporting groups
Arm/Group | Patient Navigation | Usual Care | Total
Number analyzed (Participants) | 53 | 49 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 49 | 102
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 102
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 50 | 45 | 95
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 6 | 8
  White | 45 | 40 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 53 | 49 | 102
Location [Count of Participants; unit: Participants]
  Utah | 24 | 21 | 45
  Pennsylvania | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use Disorder (OUD) and Other Substance Use Disorder (SUD) Treatment Linkage/Retention
Description: Percentage of days of days of attending outpatient and inpatient Substance Use Disorder treatment.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Control | Patient Navigation
Number analyzed (Participants) | 49 | 52
Percentage of days | -1.5 (50.2) | -8.8 (46.7)

2. Primary Outcome: Adherence to Medication-Assisted Treatment (MAT) Medication Use Section
Description: Adherence to MAT will be assessed through the treatment services review (TSR-6) medication use section defined by percentage days of attendance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage of days of attendance
Arm/Group | Control | Patient Navigation
Number analyzed (Participants) | 49 | 52
Percentage of days of attendance | 30.7 (43.8) | 40.4 (53.6)

3. Secondary Outcome: Adequacy of Prenatal Care
Description: Capturing prenatal care will be accessed through the adequacy of prenatal care utilization index (APNCU). This index will be used to determine the sufficiency of prenatal care participants received.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Patient Navigation
Number analyzed (Participants) | 43 | 49
Participants
  Adequate plus | 10 | 12
  Adequate | 13 | 15
  Intermediate | 11 | 11
  Inadequate | 9 | 11

ADVERSE EVENTS:
Time Frame: Death was the only adverse event collected.
Description: Adverse event collection started at baseline and ended at 6 months post-partum.
Arm/Group | Control | Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/49 | 1/53
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/53
Other Adverse Events (participants affected / at risk) | 0/49 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/45/NCT03833245/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03833245/ICF_001.pdf